CLINICAL TRIAL: NCT05515302
Title: Effect of Playing an Audio Clip for Pain and Anxiety Control for Burn Patients While Dressing Burn Wounds: Randomized Controlled Trial
Brief Title: Effect of Playing an Audio Clip for Pain and Anxiety Control in Patients While Dressing Burn Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Resmi Lekhadevi, Principal Investigator, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MRC-01-22-239
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Pain; Anxiety
Keywords: pain; anxiety; Burns Patients; Wound Dressing.
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: open label Randomized controlled trial
Masking Description: None are masked in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group consists of 50 Participants as per the inclusion criteria. The Audio clips will be administered to the experimental group.
  Interventions: Other: Audio Clip
- Control Group (No Intervention): The control group will not receive the intervention but will receive treatment as usual.

INTERVENTIONS:
Other: Audio Clip — Selected Audio clips will be introduced to the study subjects during the Burns Dressing Changes. The Audio Clips will be selected as per subjects preference.
  Arms: Experimental Group

SUMMARY:
The aim of this clinical trial is to assess the effect of playing patient preferred audio clip for controlling the pain and anxiety in patients while dressing burn wounds. The age group to be selected for this explicit examination is 18 years and above. The researcher will assess the pain and anxiety levels in both experimental and control groups having sample size of 50 each using standardized tools. The patient in intervention group will be offered selected audio clips to choose from. The patient preferred audio clips will be played for 10 days while the control group will be provided with treatment as usual. After collecting the data from both groups, it will be compared to analyze the effectiveness of listening to the audio clips chosen by the patient.

DETAILED DESCRIPTION:
Burn related pain and anxiety is an important health problem. Surgical procedures and physical rehabilitation is commonly associated with pain and anxiety among burn injuries. Burn pain initially associated with size and degree of burn followed by post rehabilitation procedures and infections. Pain during burn incident and expectation of pain in treatment procedures create severe anxiety in most of the patients. In this investigation researcher is going to use listening to an audio clip (piece of self-selected music, sound from nature, or religious recitations) as a non-pharmacological intervention. Audio pieces are used for clinical purposes as complementary and alternative medicine. Although it is not practiced extensively due to the lack of evidence-based results in this particular area of research. This is an open label Randomized controlled trial aimed to assess the effectiveness of listening to an audio clip as an adjunct to TAU among hospitalized burns patient.

This study is open label, prospective, parallel group, randomized control design. The trial compares thosepatients with intervention group and control group with treatment as usual. Based on the inclusion criteria those patients with 10-30% of burns and need to stay in hospital for 10 days and withpain score of >=4 will be included in the study. The samples will be divided into two groups by randomly assigning the patients to each group. The analysis will be conducted to assess the effectiveness of listening to an audio clip for controlling pain and anxiety. No blinding or masking will be performed in this study.The patients in the intervention group will be introduced to the music player before and the procedure. After the preparation of the intervention subsequently on the same day or during the next day's prior to dressing NRS and BAI will be administered to evaluate the patient's pain and anxiety levels. After completion of intervention pain, anxiety and hemodynamic parameters will be collected. Treatment as usual will be provided for all control group patients as per Unit Protocol. The primary outcome was reduced pain and anxiety levels during the dressing changes as evidenced by reducing 15-20% in experimental group as compared to control group with treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18 years and above.
* Fit the diagnostic standard of severe burn injury as per the clinical guidelines with burns up to10%
* 30% the total body surface area. (TBSA).
* Hospitalized burn patients with an expected stay in hospital for 10 days at the time of signing the informed consent.
* Patient needs to be literate to understand the instruction and the audio clip and provide response for the questionnaire.
* Pain score before intervention >=4 NRS (moderate pain

Exclusion Criteria:

* Burn patients who are critically ill with ventilator support,
* Burn patient with respiratory problem or hearing impairment,
* Burn patients with cognitive impairments.
* Burn patient with diabetic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
change in pain intensity | Throughout study completion up to 10 days after randomization.
  Measures the changes in pain intensity with a Numerical Rating Scale from 0-10 with higher score indicates higher levels of pain and lower scores indicates less pain 15-20% in experimental group as compared to control group with treatment as usual.
changes in anxiety level | Throughout study completion up to10 days after randomization.
  Measures the changes in anxiety with Beck Anxiety Inventory scale from 0-63 maximum scores. Higher scores indicate higher levels of anxiety and lower scores indicates lower levels of anxiety.

SECONDARY OUTCOMES:
changes in Heart rate | Throughout study completion up to10 days after randamization .
  Measures changes in heart rate via hospital monitors , these changes are in beats per minute(bpm) and will be obtained prior to pre-intervention phase and immediately after post intervention phase.
changes in Respiratory rate | Throughout study completion up to10 days after randomization.
  Measures changes in heart rate via hospital monitors ,these changes are in breaths per minute(bpm) and will be obtained prior to pre-intervention phase and immediately after post intervention phase.
Changes in Blood Pressure | Throughout study completion up to 10 days after randomization.
  Measures changes in blood pressure via hospital monitors ,these changes are in millimeters of mercury (mm hg) and will be obtained prior to pre-intervention phase and immediately after post intervention phase.

OTHER OUTCOMES:
Medication intake | Throughout study completion up to 10 days after randomization.
  Rescue doses asked by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
The Study data of Participants will not be shared outside Hamad Medical Corporation. The Data Will be managed according to the Norms of HMC- Medical Research Centre.